CLINICAL TRIAL: NCT00340002
Title: Fetal Anatomy by Three-Dimensional Ultrasound
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997065; OH97-CH-N065
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth; Pregnancy; Fetal Growth Abnormalities
Keywords: Fetal Anatomy; Pregnancy; Prenatal Diagnosis; Natural History
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women aged 18 years and older

SUMMARY:
A major goal of perinatal care is to accurately diagnose fetal anomalies prior to birth. This capability allows clinicians to make prudent decisions regarding antepartum care, delivery site, and postnatal therapy. Three-dimensional ultrasound is a recent technology that provides a new way to evaluate the fetus. This technique allows one to scan through a digital ultrasound volume dataset, visualize organs from different perspectives, measure volumes, and render anatomical features through computer processing. However, the accurate characterization of fetal anomalies by this technique must be interpreted in relation to normal fetal anatomy at different stages of pregnancy.

We are continuing to develop an image reference library of fetal anatomy by identifying key diagnostic features by three-dimensional ultrasound. A cross-sectional observational study of up to 1,400 fetuses will catalog a broad spectrum of congenital malformations at various gestational ages. The protocol will include up to 400 examples of normal fetal anatomy by three-dimensional ultrasonography.

All cases will be placed into a digital image database. For each anomaly category, volume reconstructions will be compared to normal anatomy at specific gestational ages. Key diagnostic findings will be documented and correlated with postnatal outcome. We anticipate that our results will permit improved diagnostic interpretation of congenital defects throughout pregnancy.

DETAILED DESCRIPTION:
A major goal of perinatal care is to accurately diagnose fetal anomalies prior to birth. This capability allows clinicians to make prudent decisions regarding antepartum care, delivery site, and postnatal therapy. Three-dimensional ultrasound is a recent technology that provides a new way to evaluate the fetus. This technique allows one to scan through a digital ultrasound volume dataset, visualize organs from different perspectives, measure volumes, and render anatomical features through computer processing. However, the accurate characterization of fetal anomalies by this technique must be interpreted in relation to normal fetal anatomy at different stages of pregnancy.

We are continuing to develop an image reference library of fetal anatomy by identifying key diagnostic features by three-dimensional ultrasound. A cross-sectional observational study of up to 7,000 fetuses will catalog a broad spectrum of congenital malformations at various gestational ages. A subset of the fetuses enrolled in this protocol will also be examined by Magnetic Resonance Imaging (MRI) to identify potential advantages and limitations of this imaging modality when compared to 3DUS for the diagnosis of congenital anomalies. The protocol will include up to 400 examples of normal fetal anatomy by three-dimensional ultrasonography.

All cases will be placed into a digital image database. For each anomaly category, volume data will be acquired at specific gestational ages. Key diagnostic features will be documented and correlated with postnatal outcome. Postnatal correlative studies may include ultrasound, MRI, X-ray, computerized tomography (CT), and photography. We anticipate that our results will permit improved diagnostic interpretation of congenital defects throughout pregnancy.

ELIGIBILITY:
* INCLUSION CRITERIA:

All pregnant subjects will be recruited under informed consent at either Hutzel or William Beaumont Hospitals.

The study population for both arms of this protocol will involve pregnant women greater than or equal to 15 years.

CROSS-SECTIONAL ARM OF PROTOCOL - NORMAL FETUS SUBJECTS:

3DUS STUDIES:

No fetal anomalies suspected by 2DUS.

Excellent visualization of normal fetal anatomy by 2DUS.

Accurate dating criteria by 1st trimester scan and/or menstrual history.

FETAL MRI STUDIES:

Gestational age between 18-42 menstrual weeks.

No known fetal abnormalities.

CROSS-SECTIONAL ARM OF PROTOCOL - ABNORMAL FETUSES:

3DUS STUDIES:

Congenital anomaly suspected by 2DUS.

Accurate dating criteria by 1st trimester scan and/or menstrual history.

FETAL MRI STUDIES:

Gestational age between 18-42 menstrual weeks.

Suspected fetal abnormalities.

POSTMORTEM STUDIES:

Suspected fetal abnormalities by prenatal ultrasound.

EXCLUSION CRITERIA:

CROSS-SECTIONAL ARM OF PROTOCOL - NORMAL FETUS SUBJECTS:

3DUS STUDIES:

Poor visualization of the fetus due to technical factors (e.g. obesity, surgical scar).

History of noncompliance with prenatal visits with the current or prior pregnancy.

FETAL MRI STUDIES:

Inability of the patient to fit in bore of MRI system.

Metallic implants that would increase risk to patient.

Previous occupational exposure to metal shop.

History of claustrophobia.

CROSS-SECTIONAL ARM OF PROTOCOL - ABNORMAL FETUSES:

3DUS STUDIES:

Poor fetal visualization from technical factors (e.g. obesity or decreased amniotic fluid).

FETAL MRI STUDIES:

Inability of the patient to fit in bore of MRI system.

Metallic implants that would increase risk to patient.

Previous occupational exposure to metal shop.

History of claustrophobia.

POSTMORTEM STUDIES:

Refusal to sign informed consent for postmortem imaging studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending Detroit Medical Center prenatal clinics in Detroit.
Sampling Method: Non-Probability Sample
Enrollment: 3650 (Actual)
Dates: Start 1997-11-26; Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Fetal Anatomy | Ongoing
  Data analysis is ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Hutzel Women's Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

REFERENCES:
- [Background] Kuo HC, Chang FM, Wu CH, Yao BL, Liu CH. The primary application of three-dimensional ultrasonography in obstetrics. Am J Obstet Gynecol. 1992 Mar;166(3):880-6. doi: 10.1016/0002-9378(92)91355-e. PMID 1550157
- [Background] Lee A, Deutinger J, Bernaschek G. "Voluvision": three-dimensional ultrasonography of fetal malformations. Am J Obstet Gynecol. 1994 May;170(5 Pt 1):1312-4. doi: 10.1016/s0002-9378(94)70148-2. PMID 8178859
- [Background] Steiner H, Staudach A, Spitzer D, Schaffer H. Three-dimensional ultrasound in obstetrics and gynaecology: technique, possibilities and limitations. Hum Reprod. 1994 Sep;9(9):1773-8. doi: 10.1093/oxfordjournals.humrep.a138793. PMID 7836537